CLINICAL TRIAL: NCT03678727
Title: Effects of Exercise on VLDL-TG Metabolism in Individuals With NAFL and NASH
Brief Title: Effects of Exercise on VLDL-TG Metabolism
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Jeyanproject2
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: NAFLD - Nonalcoholic Fatty Liver Disease; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) covers a spectrum from reversible hepatic steatosis to inflammation and fibrosis termed steatohepatitis (NASH) and cirrhosis. New evidence indicates that NAFLD is associated with development of heart failure, abnormal ventricular glucose and fatty acid (FA) utilisation and cardiosteatosis. The mechanisms behind cardiac involvement and the progression from NAFL to NASH are poorly understood but must include altered cardiac and intrahepatic lipid handling. In collaboration with renowned research groups from Oxford, Mayo Clinic and Copenhagen we plan comprehensive kinetic studies of heart and liver FA uptake and oxidation, ventricular function and substrate utilisation, and hepatic triglyceride (TG) secretion in order to assess mechanisms governing cardiac and hepatic lipid and glucose trafficking in subjects with NAFL and NASH and the relationship with heart function. In addition, we will assess skeletal muscle and adipose tissue enzyme activities, gene expression and protein concentrations in these subjects to define mechanisms involved in the cross-talk between heart, liver, muscle and adipose tissues. We will address these questions using innovative tracer techniques (11Cpalmitate, 11C acetate, 18FDG glucose PET tracers and TG tracers) in combination with hepatic vein catherisation to study cardiac and liver substrate trafficking, as well as NMR spectroscopy, echocardiography, muscle and fat biopsies in combination with state-of-the art muscle and adipose tissue enzyme kinetics, gene- and protein expression. Effects of acute exercise as well as GLP-1 agonist and SGLT-2 inhibitor treatment (alone and in combination) will be assessed. The overarching goals are to define abnormalities and differences between NAFLD and NASH in hepatic lipid (FA and TG) metabolism and to assess hepatic, adipose and skeletal muscle lipid and substrate utilisation.

ELIGIBILITY:
Inclusion Criteria:

* • 8 obese subject men with NAFL (MR spectroskopi, fibro scanner) (BMI > 30).

  * 8 obese subject men with NASH (MR spectroskopi, fibro scanner) (BMI > 30).
  * age between 40-70 years Written consent before the start of the study

Exclusion Criteria:

* known current disease
* Fixed medical drug consumption except antihypertensive drugs and statins. However, pause statins 3 weeks before the examination date
* Blood donation within the last 3 months prior to the study
* Participation in experiments involving radioactive isotopes within the last 3 months
* Alcohol abuse (over 21 items per week for men and 14 for women)
* Smoking
* Weight over 130 kg
* Cancer patients
* Large intake of medication

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 8 obese subject men with NAFL (MR spectroskopi, fibro scanner) (BMI > 30). 8 obese subject men with NASH (MR spectroskopi, fibro scanner) (BMI > 30).
  • age between 40-70 years Written consent before the start of the study
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Effects of exercise on VLDL-TG metabolism in individuals with NAFL or NASH | 3 years
  * VLDL-TG turnover (µmol/min)
  * To evaluate the acute effects of exercise on VLDL-TG secretion and clearance
  * To assess the uptake and cellular/intracellular regulation of FFA and VLDL-TG in fat and muscle tissue
Effects of exercise on VLDL-TG metabolism in individuals with NAFL or NASH | 3 years
  LPL-activity (µmol/time)

SECONDARY OUTCOMES:
Compare the acute effects of exercise in individuals with NAFL or NASH | 3 years
  Oxidation of VLDL-TG-FA(µmol/min)
Compare the acute effects of exercise in individuals with NAFL or NASH | 3 years
  FFA turnover (µmol/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Arhus University Hospital Department of Endocrinology and Internal Medicine, Skejby, Aarhus N, Denmark